CLINICAL TRIAL: NCT03076073
Title: Ultrasonography of the Patellar Tendon and Achilles Tendon in Children Adolescent and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dan Nemet, MD, Prof. Dan Nemet, Meir Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MeirMc0321-16CTIL
Record Dates: First submitted 2017-03-05; First posted 2017-03-09 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Obesity, Childhood; Obesity; Tendon Thickening
Keywords: Ultrasound; Achilles tendon; Patellar tendon; obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluating Tendons Structures (No Intervention): Ultrasound measurements of Patellar Tendon and Achilles Tendon Structures
- Impact of physical activity on tendons (Active Comparator): Ultrasound measurements of Patellar Tendon and Achilles Tendon Structures following different types and different intensity of physical activity
  Interventions: Other: Impact of physical activity on tendons

INTERVENTIONS:
Other: Impact of physical activity on tendons — Single vs. multiple (up to 12 weeks) of different types of physical exercises (aerobic vs. anaerobic activities).
  Arms: Impact of physical activity on tendons

SUMMARY:
The aim of the current study is to evaluate the Patellar tendon and Achilles tendon structures among children, adolescents and adults with different weight status. That in order to improve our understanding on the impact of acute and overused loads on tendon structure; and, in developing strategies to reduce tendon's injuries following physical exercises.

DETAILED DESCRIPTION:
Studies showed that the probability of tendon abnormalities is higher in obese subjects compared to normal weight peer. Adiposity has been recognized as a risk factor for alterations in load- bearing tendons; and, different impact of loading exercises on tendon structure has been reported for obese individuals compared to normal weight individuals. The aim of the current study is to evaluate the Patellar tendon and Achilles tendon structures among children, adolescents and adults with different weight status. That in order to improve our understanding on the impact of acute and overused loads on tendon structure; and, in developing strategies to reduce tendon's injuries following physical exercises.

Tendon structure would be evaluated with UTC-imaging ultrasound device. UTC imaging allows for three-dimensional imaging of the tendon, semi- quantification of structure, and calculation of tendon dimensions. The resultant UTC analysis quantify the tendon into four echo types (I-IV) based on the stability of pixel brightness over contiguous images allowing inferences to be made on the alignment of tendon bundles. Briefly, echo types I and II correspond with relatively high stability in gray-scale pixel brightness over contiguous images due to one resulting US signal transmission. These echo types correspond with aligned fibrillar structure (AFS) within the tendon. Echo types III and IV are generated by multiple signal transmission that interfere as a consequence of multiple interfaces. These echo types represent a disorganized amorphous fibrillar structure that has non parallel ﬁber arrangement. For this study, the relative percentage and (muscle cross section area (mCSA) of these parameters were the main outcomes investigated. A linear-array US transducer (SmartProbe, A 10- megahertz (MHz) linear-array transducer, USA) mounted within a customized tracking device with motor drive and built-in acoustic stand off pad (UTC Tracker, UTC Imaging, Netherlands) was placed on the skin, perpendicular to the long axis of the tendon (Achilles or patellar), ensuring that the calcaneus or inferior pole of the patella was visible. Coupling gel was applied between the transducer, standoff pad, and skin to ensure maximum contact. Once a clear transverse image of the tendon and bony landmark was established, the motor drive automatically moved the transducer over the length of the tendon capturing a transverse grayscale US image every 0.2 mm over a distance of 12 cm. By compounding these images, a gray-scale US image data block is rendered that allows the tendon to be viewed in three planes: transverse, sagittal, and coronal (UTC2010, UTC Imaging). From this data block, each tendon was classified as either normal or pathological.

Each participant would be measured at both Achilles tendons and both Patellar tendons (total time 10min) while prone position (for the Achilles tendon) and in sitting position (for Patellar tendon). Each screening is for 45sec.

* Participants in different ages and different weight status would be measured for tendon structure
* Tendon structure would be evaluated following single and multiple (up to 12 weeks) aerobic and anaerobic exercises.

ELIGIBILITY:
Inclusion Criteria: - participants should be between the ages of 6 to 30 years; normal-weight, over-weight and obese participants.

Exclusion Criteria:

* participants that had orthopedic surgery or professional athletes.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Ultrasound tissue characterization | 10min
  Based on the stability of echo-pattern the device can discriminate 4 different echo-types of tendon specimen

SECONDARY OUTCOMES:
Ultrasound 3-D visualization of tendon structure | 10min
  measuring the total volume of the tendon; anterior-posterior and medial-lateral diameters

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, Prof., Principal Investigator — Meir Medical Center
Locations (1):
- 'Meir children's sport and health center', Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No